CLINICAL TRIAL: NCT05457452
Title: Comparison of Functional Outcomes in Patients Using Knee Brace and Without Knee Brace After Anterior Cruciate Ligament Reconstruction Surgery With Autograft Bone Quadricep Tendon Arthroscopy
Brief Title: Functional Outcomes Comparison in Patients Using Knee Brace Post ACL Reconstruction With Autograft Bone Quadricep Tendon
Acronym: ACL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Danarto Hari Adhimukti, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INDO321
Record Dates: First submitted 2022-07-02; First posted 2022-07-14 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Anterior Cruciate Ligament Injuries; Arthroscopy; Braces
Keywords: Anterior Cruciate Ligament Injuries; Arthroscopy; Knee Braces; Functional Outcome
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Intervention Model Description: All patients at Cipto Mangunkusumo Hospital and Gatot Soebroto Hospital, who underwent ACL reconstruction in the period January 2022 - January 2022 who met the inclusion and exclusion criteria.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Knee Brace (Experimental): Use of a Knee Brace after ACL Reconstruction, the patient is put on a knee brace by an orthopedic doctor or orthopedic resident after ACL reconstruction
  Interventions: Device: Knee Brace
- No Knee Brace (No Intervention)

INTERVENTIONS:
Device: Knee Brace — Installation of an angle-adjustable knee brace, used after ACL reconstruction performed by an orthopedic specialist or orthopedic PPDS with the first week the angle locked at 00, in the second week the angle 0-900, in the third week the angle 0-1200, and the fourth week the angle of flexion full. Braces are used except for physical therapy according to the rehabilitation protocol in the first week.
  Arms: Knee Brace

SUMMARY:
This study is a study looking for the relationship between variables with a prospective cohort design to determine functional outcomes subjectively and objectively in patients with and without braces after ACL reconstruction with bone quadriceps tendon per arthroscopy.

DETAILED DESCRIPTION:
This study is a study looking for the relationship between variables with a prospective cohort design to determine functional outcomes subjectively and objectively in patients with and without braces after ACL reconstruction with bone quadriceps tendon per arthroscopy.

The research will be conducted at the National Central General Hospital dr. Cipto Mangunkusumo, Jakarta Police Hospital and Gatot Soebroto Army Hospital in Jakarta, Indonesia.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with age more than equal to 18 years
* Patients with ACL rupture without other ligament ruptures undergoing ACL reconstruction
* Patients undergoing ACL reconstruction using Quadricep Tendon Autograft

Exclusion Criteria:

* Patients with hyperlaxity
* Patients with previous history of ACL reconstruction
* Patients with recurrent rupture during the observation period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
International Knee Documentation Committee (IKDC) score 3 months post treatment | 3 months
  Patients were interviewed by the examiner based on questions in the International Knee Documentation Committee (IKDC) form. Scale from 0 to 100. Higher score means better clinical outcomes
International Knee Documentation Committee (IKDC) score 6 months post treatment | 6 months
  Patients were interviewed by the examiner based on questions in the International Knee Documentation Committee (IKDC) form. Scale from 0 to 100. Higher score means better clinical outcomes
Lysholm score 3 months post treatment | 3 months
  Patients were interviewed by the examiner based on the questions in the Lysholm form. Scale from 0 to 100. Higher score means better clinical outcomes
Lysholm score 6 months post treatment | 6 months
  Patients were interviewed by the examiner based on the questions in the Lysholm form. Scale from 0 to 100. Higher score means better clinical outcomes
Knee injury and Osteoarthritis Outcome (KOOS) score 3 months post treatment | 3 months
  The patient was interviewed by the examiner according to the KOOS Questionnaire form. Scale from 0 to 100. Higher score means better clinical outcomes
Knee injury and Osteoarthritis Outcome (KOOS) score 6 months post treatment | 6 months
  The patient was interviewed by the examiner according to the KOOS Questionnaire form. Scale from 0 to 100. Higher score means better clinical outcomes
Anterior Cruciate Ligament Return to Sport after Injury (ACL-RSI) score 3 months post treatment | 3 months
  Patients were interviewed by the examiner based on the questions on the Anterior Cruciate Ligament Return to Sport After Injury (ACL-RSI) form. Scale from 0 to 100. Higher score means better clinical outcomes
Anterior Cruciate Ligament Return to Sport after Injury (ACL-RSI) score 6 months post treatment | 6 months
  Patients were interviewed by the examiner based on the questions on the Anterior Cruciate Ligament Return to Sport After Injury (ACL-RSI) form. Scale from 0 to 100. Higher score means better clinical outcomes
Rolimeter 3 months post treatment | 3 months
  Objective examination of knee stability using a rolymeter
Rolimeter 6 months post treatment | 6 month
  Objective examination of knee stability using a rolymeter

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Orthpaedic and Traumatology RSCM-FKUI, Jakarta Pusat, Jakarta Special Capital Region, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lowe WR, Warth RJ, Davis EP, Bailey L. Functional Bracing After Anterior Cruciate Ligament Reconstruction: A Systematic Review. J Am Acad Orthop Surg. 2017 Mar;25(3):239-249. doi: 10.5435/JAAOS-D-15-00710. PMID 28195986
- [Background] Kaeding CC, Leger-St-Jean B, Magnussen RA. Epidemiology and Diagnosis of Anterior Cruciate Ligament Injuries. Clin Sports Med. 2017 Jan;36(1):1-8. doi: 10.1016/j.csm.2016.08.001. Epub 2016 Oct 4. PMID 27871652
- [Background] Montalvo AM, Schneider DK, Webster KE, Yut L, Galloway MT, Heidt RS Jr, Kaeding CC, Kremcheck TE, Magnussen RA, Parikh SN, Stanfield DT, Wall EJ, Myer GD. Anterior Cruciate Ligament Injury Risk in Sport: A Systematic Review and Meta-Analysis of Injury Incidence by Sex and Sport Classification. J Athl Train. 2019 May;54(5):472-482. doi: 10.4085/1062-6050-407-16. Epub 2019 Apr 22. PMID 31009238
- [Background] Chan CX, Wong KL, Toh SJ, Krishna L. Epidemiology of patients with anterior cruciate ligament injuries undergoing reconstruction surgery in a multi-ethnic Asian population. Res Sports Med. 2021 Jan-Feb;29(1):12-24. doi: 10.1080/15438627.2018.1492391. Epub 2018 Jul 9. PMID 29985059
- [Background] Dzakiya FNA, Tinduh D, Utomo DN. Risk Estimation of Anterior Cruciate Ligament (ACL) Injury in East Java Puslatda Pencak Silat Athletes. Surabaya Phys Med Rehabil J. 2021;3:29.
- [Background] Lubis AM, Dasril DF. Comparison of functional outcome between bone quadriceps tendon (BQT) and single-bundle hamstring tendon (SBHT) autograft in arthroscopic-assisted anterior cruciate ligament reconstruction cases: a prospective cohort study. Ann Med Surg (Lond). 2020 Nov 13;60:509-514. doi: 10.1016/j.amsu.2020.11.023. eCollection 2020 Dec. PMID 33294183
- [Background] Rudy, Mustamsir E, Phatama KY. Tensile strength comparison between peroneus longus and hamstring tendons: A biomechanical study. Int J Surg Open [Internet]. 2017;9:41-4. Available from: https://doi.org/10.1016/j.ijso.2017.10.002
- [Background] Fleming BC, Renstrom PA, Beynnon BD, Engstrom B, Peura G. The influence of functional knee bracing on the anterior cruciate ligament strain biomechanics in weightbearing and nonweightbearing knees. Am J Sports Med. 2000 Nov-Dec;28(6):815-24. doi: 10.1177/03635465000280060901. PMID 11101104
- [Background] Perrone GS, Webster KE, Imbriaco C, Portilla GM, Vairagade A, Murray MM, Kiapour AM. Risk of Secondary ACL Injury in Adolescents Prescribed Functional Bracing After ACL Reconstruction. Orthop J Sports Med. 2019 Nov 12;7(11):2325967119879880. doi: 10.1177/2325967119879880. eCollection 2019 Nov. PMID 31763340
- [Background] Melegati G, Tornese D, Bandi M, Volpi P, Schonhuber H, Denti M. The role of the rehabilitation brace in restoring knee extension after anterior cruciate ligament reconstruction: a prospective controlled study. Knee Surg Sports Traumatol Arthrosc. 2003 Sep;11(5):322-6. doi: 10.1007/s00167-003-0386-3. Epub 2003 Jul 16. PMID 12879225